CLINICAL TRIAL: NCT06717113
Title: Clinical PET Imaging Evaluation of 68Ga-BC1 Probe in Multiple Myeloma
Brief Title: A Molecular Probe Targeting BCMA for the Clinical Diagnosis of Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Tianyao Wang, Principal Investigator, Peking University First Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUFH-MM-BC1
Record Dates: First submitted 2024-09-28; First posted 2024-12-04 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma and Malignant Plasma Cell Neoplasms
Keywords: multiple myeloma; molecular probe; Immuno-PET
MeSH Terms: conditions — Multiple Myeloma | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: This study is an interventional clinical trial in which enrolled patients will undergo a comparative analysis using two PET/CT imaging agents: 68Ga-NB381 and 18F-FDG. The two drugs should be given at least one day apart.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 68Ga-BC1 PET/CT diagnosis (Experimental)
  Interventions: Drug: 68Ga-BC1
- 18F-FDG PET/CT diagnosis (Active Comparator)
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — Prior to the examination, patients will be required to fast for at least 6 hours. 18F-FDG (0.05-0.1 mCi/kg) will be intravenously injected, and one hour after the injection, head and torso imaging will be performed using a Shanghai United Imaging uMI 780 PET/CT scanner, covering the region from the top of the head to the upper third of the thigh. The patient will lie supine and breathe calmly during the procedure. After image acquisition, the data will be reconstructed using the OSEM method to generate coronal, sagittal, transverse, and PET/CT fusion images.
  Arms: 18F-FDG PET/CT diagnosis
Drug: 68Ga-BC1 — The prepared and quality-controlled 68Ga-BC1 (0.05-0.1 mCi/kg) will be intravenously injected into the patient. Two hours after the injection, whole-body imaging will be performed using a Shanghai United Imaging uMI 780 PET/CT scanner, covering the region from the top of the head to the mid-thigh. If any indeterminate lesions are found during the routine imaging, delayed imaging will be performed for further differentiation. The patient will lie supine and breathe calmly during the procedure. After image acquisition, the data will be reconstructed using the OSEM method to generate coronal, sagittal, transverse, and PET/CT fusion images.
  Arms: 68Ga-BC1 PET/CT diagnosis

SUMMARY:
Multiple Myeloma (MM), the second most common hematological malignancy, continues to pose challenges in precise clinical identification. As a potential solution, nuclear medicine immuno-PET imaging has emerged as a promising approach. However, traditional full-length antibody probes suffer from delayed tumor uptake peaks and low target-to-background ratios, limiting their clinical utility. In our study, a peptide or nanobody targeting BCMA was developed by computer-aided designing, which was subsequently radiolabeled with 68Ga to create a novel molecular probe, 68Ga-MM-BC1. This research aims to overcome the diagnostic limitations of MM and may also offer valuable insights for molecular-targeted imaging in other malignant tumors.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) predominantly affects the elderly and often presents insidiously, with most patients being diagnosed at an advanced stage. As China's population ages, the incidence of MM is increasing, now surpassing that of acute leukemia. The primary clinical manifestation is bone destruction, which lacks specificity. Diagnosis primarily relies on invasive bone marrow biopsies to detect clonal plasma cell proliferation. However, improper selection of the biopsy site can lead to false-negative results. BCMA is highly expressed on the surface of malignant plasma cells in MM, making it a characteristic tumor biomarker for this disease.

With the rising incidence of malignant tumors in China, there is an increasing demand for radiopharmaceuticals in clinical practice. Given the limitations of 18F-FDG in PET imaging, particularly regarding specificity, the development of novel targeted nuclear medicine molecular probes holds significant academic and clinical value. This is especially true for monitoring the therapeutic effects of peptide or nanobody-based treatments targeting BCMA, which offers distinct advantages. This project focuses on utilizing a peptide or nanobody with high affinity for BCMA as the targeting group for radiopharmaceuticals, exploring the diagnostic efficacy of 68Ga-BC1 in MM patients with high BCMA expression. This approach not only aids in the early diagnosis of MM but also helps tailor effective precision treatments for patients based on their BCMA expression levels.

68Ga-BC1, a novel BCMA-targeting molecular probe labeled with 68Ga, has potential applications in the diagnosis and research of various BCMA-expressing malignancies, including MM. 68Ga-BC1 is synthesized using THP as a bifunctional chelator to coordinate with 68Ga^3+, and the labelling process is simple, allowing for direct use without purification. It demonstrates high in vivo stability and significant tumor uptake in tumor-bearing mice, with superior imaging performance. In this project, the automated labelling process of 68Ga-BC1 will be studied, and quality control measures for the resulting radiopharmaceutical injection will be established. A quality standard for this new PET probe will be set, laying the groundwork for the clinical translation of this drug within China. This study aims to provide valuable data on 68Ga-BC1 PET/CT imaging, offering insights for the early diagnosis, treatment planning, and efficacy evaluation of patients with BCMA-expressing malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Suspected multiple myeloma patients scheduled for bone marrow aspiration or tissue biopsy within the past 3 months; able to fully understand and voluntarily participate in the study, with signed informed consent; able to cooperate with the examination.
* Diagnosed symptomatic multiple myeloma patients; able to fully understand and voluntarily participate in the study, with signed informed consent; able to cooperate with the examination.

Exclusion Criteria:

* Pregnant women; individuals unable to understand the examination process or who are unable to cooperate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
MM patients will be recruited to undergo PET/CT imaging using 68Ga-NB381 and 18F-FDG to evaluate and verify that the imaging agent 68Ga-NB381 can safely and effectively identify lesions. | All PET/CT images will be reviewed by physicians, and a unified diagnostic opinion will be provided within 3 days after adminis. After imaging, patients will be scheduled for follow-up visits every 3 months, with a follow-up period of at least 12 months.
  This study will investigate the radioactive uptake of 68Ga-BC1 in lesion sites of multiple myeloma patients and evaluate the ability of 68Ga-BC1 to detect BCMA overexpression in these patients.
  According to the admission and exclusion criteria, patients who meet the conditions are screened. After the patients were enrolled, baseline examination information was collected, including blood routine, blood biochemistry, tumour markers, histopathological diagnosis results, imaging diagnosis results, etc.
  For the Follow-up information, the patient's bone marrow aspirate or pathological tissue biopsy, laboratory test results (blood monoclonal M protein, 24-hour urine light chain, etc.), bone scintigraphy, CT or MR and other imaging examination results would be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Kang, M.D., Study Chair — Peking University First Hospital; Yujun Dong Dong, M.D., Study Director — Peking University First Hospital; Tianyao Wang, Ph.D., Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Department of Nuclear Medicine, Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
Some representative clinical trial results will be used for publication in ICMJE journals.
Supporting Information: CSR
Time Frame: January 2025-December 2027
Access Criteria: The ICMJE journals and their readers.

REFERENCES:
- [Background] Kang L, Jiang D, England CG, Barnhart TE, Yu B, Rosenkrans ZT, Wang R, Engle JW, Xu X, Huang P, Cai W. ImmunoPET imaging of CD38 in murine lymphoma models using 89Zr-labeled daratumumab. Eur J Nucl Med Mol Imaging. 2018 Jul;45(8):1372-1381. doi: 10.1007/s00259-018-3941-3. Epub 2018 Feb 15. PMID 29450576
- [Background] Kang L, Li C, Rosenkrans ZT, Engle JW, Wang R, Jiang D, Xu X, Cai W. Noninvasive Evaluation of CD20 Expression Using 64Cu-Labeled F(ab')2 Fragments of Obinutuzumab in Lymphoma. J Nucl Med. 2021 Mar;62(3):372-378. doi: 10.2967/jnumed.120.246595. Epub 2020 Aug 21. PMID 32826320
- [Background] Kang L, Li C, Yang Q, Sutherlin L, Wang L, Chen Z, Becker KV, Huo N, Qiu Y, Engle JW, Wang R, He C, Jiang D, Xu X, Cai W. 64Cu-labeled daratumumab F(ab')2 fragment enables early visualization of CD38-positive lymphoma. Eur J Nucl Med Mol Imaging. 2022 Apr;49(5):1470-1481. doi: 10.1007/s00259-021-05593-9. Epub 2021 Oct 22. PMID 34677626